CLINICAL TRIAL: NCT02101385
Title: A Phase II Randomized Controlled Trial of Genomically Directed Therapy After Preoperative Chemotherapy in Patients With Triple Negative Breast Cancer: Hoosier Oncology Group BRE12-158
Brief Title: Randomized Controlled Trial of Genomically Directed Therapy in Patients With Triple Negative Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bryan Schneider, MD (Other)
Collaborators: Hoosier Cancer Research Network (Other); Vera Bradley Foundation for Breast Cancer (Other); Walther Cancer Institute (Other); Indiana University (Other)
Responsible Party: Sponsor-Investigator, Bryan Schneider, MD, Sponsor-Investigator, Hoosier Cancer Research Network
Organization: Hoosier Cancer Research Network (Other)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: BRE12-158
Record Dates: First submitted 2014-03-21; First posted 2014-04-02 (Estimated); Results first posted 2023-09-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-08

CONDITIONS: Malignant Neoplasm of Breast; Breast Cancer
Keywords: Genomically-Directed Therapy; DNA Sequencing; RNA Sequencing
MeSH Terms: conditions — Breast Neoplasms | interventions — Observation; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (Genomically Directed Monotherapy) (Experimental): Participants randomized to Experimental Arm A will receive an FDA approved drug at standard dose for four cycles (12-16 weeks total duration, depending on cycle length). Clinical and laboratory monitoring and dose-reductions will follow the FDA package insert guidelines.
  Interventions: Drug: Genomically Directed Monotherapy
- Control Arm B (Observation/Standard Therapy) (Other): Currently no standard therapy has proven efficacy in this patient population and thus observation alone would be considered standard of care. Additional therapy is permitted, however, if deemed appropriate by the treating physician.
  Interventions: Other: Observation/Standard Therapy

INTERVENTIONS:
Drug: Genomically Directed Monotherapy — Participants randomized to Experimental Arm A will receive an FDA approved drug at standard dose for four cycles (12-16 weeks total duration, depending on cycle length). The CGTB will assign therapy to each participant individually based on biomarkers/pathways identified by DNA sequencing:
  Arms: Arm A (Genomically Directed Monotherapy)
Other: Observation/Standard Therapy — Currently no standard therapy has proven efficacy in this patient population and thus observation alone would be considered standard of care. Additional therapy is permitted, however, if deemed appropriate by the treating physician.
  Arms: Control Arm B (Observation/Standard Therapy)

SUMMARY:
This study will test the theory that therapy designed for each individual's tumor will improve outcomes over standard of care in a population that needs a better standard.

DETAILED DESCRIPTION:
OUTLINE: This is a multi-center trial.

SEQUENCING:

DNA from archived tumor samples collected at the time of surgery (residual disease post neoadjuvant chemotherapy) will be extracted and sequenced. The resulting sequencing data will be interrogated for known genomic drivers of sensitivity or resistance to existing FDA approved agents.

CANCER GENOMICS TUMOR BOARD (CGTB):

Realizing that optimal treatment recommendations cannot be made based on sequencing data alone, the CGTB will be responsible for the final treatment recommendation. The CGTB will consider the genomic data along with the patient's prior treatment history, ongoing toxicities, and comorbidities. Preference will be given to the treatment identified by the sequencing data unless a significant clinical or safety contraindication exists for that therapy. All participants and investigators will be blinded to sequencing results and CGTB deliberations until the time of relapse.

PARTICIPANTS WITH A CGTB TREATMENT RECOMMENDATION:

Participants with a CGTB recommendation will be randomized to Experimental Arm A (genomically directed monotherapy) or Control Arm B (standard therapy).

EXPERIMENTAL ARM A (GENOMICALLY DIRECTED MONOTHERAPY):

Participants randomized to Experimental Arm A will receive an FDA approved drug at standard dose for four cycles (12-16 weeks total duration, depending on cycle length). Clinical and laboratory monitoring and dose-reductions will follow the FDA package insert guidelines.

TOP GENOMIC ACTIONABLE BIOMARKERS/PATHWAYS AND DRUG RECOMMENDATIONS:

1. PIK3CA, PTEN: Everolimus
2. TOP2A: Doxorubicin
3. PARP1, BRCA1: Cisplatin and Olaparib
4. VEGFA: Bevacizumab
5. TYMP: Capecitabine
6. SSTR2: Octreotide
7. MGMT: Temozolomide
8. MYC: Paclitaxel
9. EGFR: Cetuximab
10. COX2: Celecoxib
11. hENT: Gemcitabine
12. MET: Crizotinib

CONTROL ARM B (STANDARD THERAPY); Recently, a randomized phase III trial of over 900 HER2-negative patients demonstrated an improvement in disease-free survival (DFS) and overall survival (OS) for the addition of 8 cycles of capecitabine in the post-neoadjuvant setting. The hazard ratios were also significant in the triple negative subgroup. Thus, capecitabine can be considered a standard option in this setting. As this represents only a single trial (with prior data not demonstrating benefit for the addition of capecitabine in the neoadjuvant nor adjuvant settings in unselected patients), observation can be considered an option as directed by the treating physician. While not recommended, other therapies can be used as deemed appropriate by the treating physician.

In the event of disease progression on the control arm, patient sequencing results will be forwarded to the treating physician.

PARTICIPANTS WITH NO CGTB RECOMMENDATION:

Participants may have no CGTB recommendation either because 1) sequencing did not identify a matched drug or 2) the matched drug was contraindicated. These participants will be assigned to Control Arm B and treated as described above for Control Arm B. As the outcome of participants without an 'actionable' genomically directed therapy may differ, the primary analysis will include only participants randomized to Control Arm B.

Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 within 14 days prior to study registration

Life Expectancy: Not Specified

Adequate laboratory values must be obtained within 14 days prior to study registration:

Hematopoietic:

* Hemoglobin (Hgb) ≥ 9.0 g/dL
* Platelets ≥ 100 K/mm3
* Absolute neutrophil count (ANC) ≥ 1.5 K/mm3

Hepatic:

* Bilirubin ≤ 1.5 x ULN (except in participants with documented Gilbert's disease, who must have a total bilirubin ≤ 3.0 mg/dL)
* Aspartate aminotransferase (AST, SGOT) ≤ 2.5 x ULN
* Alanine aminotransferase (ALT, SGPT) ≤ 2.5 x ULN

Renal:

* Calculated creatinine clearance of ≥ 50 cc/min using the Cockcroft-Gault formula

Cardiac:

* Left ventricular ejection fraction within normal limits obtained within 30 days prior to study registration. NOTE: Participants with an unstable angina or myocardial infarction within 12 months of study registration are excluded.
* No clinically significant arrhythmia or baseline ECG abnormalities in the opinion of the treating physician

ELIGIBILITY:
Inclusion Criteria:

-Written informed consent and HIPAA authorization for release of personal health information.

NOTE: HIPAA authorization may be included in the informed consent or may be obtained separately.

NOTE: Central pathology review may be conducted any time after definitive surgery. Consenting participants may be pre-registered to the study and proceed with central pathology review before full eligibility has been confirmed. However, ALL of the eligibility criteria must be met and formal study registration completed prior to submission of the sample for sequencing.

* Age ≥ 18 years at the time of consent.
* ECOG Performance Status 0 or 1 within 14 days prior to study registration.
* Women and men of childbearing potential must be willing to use an effective method of contraception (e.g. hormonal or barrier method of birth control; abstinence) from the time consent is signed until 4 weeks after protocol therapy discontinuation.
* Women of childbearing potential must have a negative pregnancy test within 30 days prior to study registration. Women should be counseled regarding acceptable birth control methods to utilize from the time of screening to start of treatment. If prior to treatment after discussion with the subject it is felt by the treating physician there is a possibility the subject is pregnant a pregnancy test should be repeated.

NOTE: Women are considered not of childbearing potential if they are surgically sterile (they have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy), or they are postmenopausal for at least 12 consecutive months.

* Women must not be breastfeeding.
* Must have histologically or cytologically confirmed triple negative (ER-/PR-/HER2-) invasive breast cancer, clinical stage I-III at diagnosis (AJCC 6th edition) based on initial evaluation by physical examination and/or breast imaging prior to study registration. NOTE: ER, PR and HER2 status will be confirmed by central pathology review prior to randomization. ER and PR will be considered negative if ≤ 1% of cells stain weakly positive. HER2 will be considered negative if scored 0 or 1+ by immunohistochemistry (IHC) or 2+ by IHC associated with a fluorescence in situ hybridization (FISH) ratio of < 2.0 or < 6 copies per cell.
* Must have completed preoperative (neoadjuvant) chemotherapy. NOTE: Acceptable preoperative regimens include an anthracycline or a taxane, or both. Participants who received preoperative therapy as part of a clinical trial may enroll. Participants may not have received adjuvant chemotherapy after surgery prior to randomization. Bisphosphonate use is allowed.
* Must have completed definitive resection of primary tumor. The most recent surgery for breast cancer must have been completed at least 14 days prior (but no more than 84 days prior) to study registration. NOTE: Negative margins for both invasive and ductal carcinoma in situ (DCIS) are desirable, however participants with positive margins may enroll if the treatment team believes no further surgery is possible and patient has received radiotherapy. Participants with margins positive for lobular carcinoma in situ (LCIS) are eligible. Either mastectomy or breast conserving surgery (including lumpectomy or partial mastectomy) is acceptable.
* Must have significant residual invasive disease at the time of definitive surgery following preoperative chemotherapy. Significant residual disease is defined as at least one of the following:

  * Residual Cancer Burden (RBC) classification II or III^6
  * Residual invasive disease in the breast measuring at least 2 cm. The presence of DCIS without invasion does not qualify as residual disease in the breast.
  * Residual invasive disease in the breast measuring at least 1cm with any lymph node involvement (does not include metastases in lymph node which are only detected by immunohistochemistry).
  * Any lymph node involvement that results in 20% cellularity or greater regardless of primary tumor site involvement (includes no residual disease in the breast).
* Must have an FFPE tumor block with tumor cellularity of 20% or greater. NOTE: Prior to randomization, the tumor cellularity will be confirmed by central pathology review and percent values will be double checked at Paradigm (a Next Generation Sequencing Company).
* BREAST RADIOTHERAPY:

  * Whole breast radiotherapy is required for participants who underwent breast-conserving therapy, including lumpectomy or partial mastectomy. Participants must have completed radiotherapy at least 14 days prior (but no more than 84 days prior) to study registration.
  * Participants with a primary tumor > 5 cm or involvement of ≥4 lymph nodes who require a mastectomy must also have radiotherapy pre- or post-operatively at the discretion of the treating physician. For participants with primary tumors ≤ 5 cm or with < 4 involved lymph nodes, provision of post-mastectomy radiotherapy is at the discretion of the treating physician. Registration must occur within 84 days of the completion of the last local therapy.
  * For radiation required prior to surgery, the participant must register within 84 days of surgery. Also, participants in this situation would not be required to have additional post-mastectomy radiation therapy.
  * For those participants who do not require radiation, registration must be within 84 days of surgery.
* No stage IV (metastatic) disease, however no specific staging studies are required in the absence of symptoms or physical exam findings that would suggest distant disease.
* No treatment with any investigational agent within 30 days prior to study registration.
* No history of chronic hepatitis B or untreated hepatitis C.
* Adequate laboratory values must be obtained within 14 days prior to study registration.

  * Hemoglobin (Hgb) >/= 9.0 g/dL
  * Platelets >/= 100 K/mm^3
  * Absolute neutrophile count (ANC) >/= 1.5 K/mm^3
  * Calculated creatinine clearance of >/= 50 cc/min using the Cockcroft-Gault formula:

    * Males: (140-Age in years) x Actual body weight in kg / 72 x Serum creatinine (mg/dL)
    * Females: Estimated creatinine clearaNCE FOR MALES X 0.85
  * Bilirubin </= 1.5 x ULN (except in participants with documented Gilbert's disease, who must have a total bilirubin </= 3.0 mg/dL)
  * Aspartate aminotransferase (AST, SGOT) </= 2.5 x ULN
  * Alanine aminotransferase (ALT, SGPT) </= 2.5 x ULN
* Left ventricular ejection fraction within normal limits obtained within 30 days prior to study registration.

NOTE: Participants with an unstable angina or myocardial infarction within 12 months of study registration are excluded.

* No clinically significant infections as judged by the treating physician.
* Must consent to allow submission of adequate archived tumor tissue sample from definitive surgery for genomic assessment of tumor.
* Must consent to collection of whole blood samples for genomic analysis
* No clinically significant arrhythmia or baseline ECG abnormalities in the opinion of the treating physician.

Exclusion Criteria:

* No stage IV (metastatic) disease, however no specific staging studies are required in the absence of symptoms or physical exam findings that would suggest distant disease.
* No treatment with any investigational agent within 30 days prior to study registration.
* No history of chronic hepatitis B or or untreated hepatitis C.
* No clinically significant infections as judged by the treating physician.
* No active second malignancy (except non-melanomatous skin cancer or incidental prostate cancer found on cystectomy): Active second malignancy is defined as a current need for cancer therapy or a high possibility (> 30%) of recurrence during the study. Previous contralateral breast cancer is allowable unless it meets "active" criteria as stated above.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 193 (Actual)
Dates: Start 2014-04-03 (Actual); Primary Completion 2021-02-21 (Actual); Study Completion 2022-09-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bryan Schneider, M.D., Study Chair — Hoosier Cancer Research Network
Locations (29):
- United States (29):
  - University of Alabama Hematology Oncology Clinic at Medical West, Birmingham, Alabama
  - Georgetown University: Lombardi Comprehensive Cancer Center, Washington D.C., District of Columbia
  - University of Florida: Shands Cancer Center, Gainesville, Florida
  - Memorial Cancer Institute, Hollywood, Florida
  - University of Miami, Sylvester Comprehensive Cancer Center, Miami, Florida
  - Memorial Breast Cancer Center: Memorial West, Pembroke Pines, Florida
  - Emory University: Winship Cancer Institute, Atlanta, Georgia
  - University of Chicago Medicine, Chicago, Illinois
  - Community Hospital of Anderson and Madison County, Inc, Anderson, Indiana
  - Fort Wayne Oncology & Hematology, Inc., Fort Wayne, Indiana
  - IU Health Goshen Hospital, Goshen, Indiana
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Community Regional Cancer Center, Indianapolis, Indiana
  - St. Vincent Hospital, Indianapolis, Indiana
  - IU Health Arnett Cancer Center, Lafayette, Indiana
  - Community Healthcare System: Monroe Medical Associates, Munster, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - Meritus Center for Clinical Research, Hagerstown, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Washington University: Siteman Cancer Center, St Louis, Missouri
  - Nebraska Cancer Specialists, Omaha, Nebraska
  - University of Cincinnati Cancer Institute, Cincinnati, Ohio
  - Mercy Clinic Oncology & Hematology: McAuley, Oklahoma City, Oklahoma
  - Pinnacle Health Cancer Center, Harrisburg, Pennsylvania
  - Erlanger Health System, Chattanooga, Tennessee
  - Joe Arrington Cancer Research and Treatment Center, Lubbock, Texas
  - Virginia Oncology Associates, Norfolk, Virginia
  - Froedtert/Medical College of Wisconsin, Milwaukee, Wisconsin
  - Aurora Health Care, Wauwatosa, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schneider BP, Jiang G, Ballinger TJ, Shen F, Chitambar C, Nanda R, Falkson C, Lynce FC, Gallagher C, Isaacs C, Blaya M, Paplomata E, Walling R, Daily K, Mahtani R, Thompson MA, Graham R, Cooper ME, Pavlick DC, Albacker LA, Gregg J, Solzak JP, Chen YH, Bales CL, Cantor E, Hancock BA, Kassem N, Helft P, O'Neil B, Storniolo AMV, Badve S, Miller KD, Radovich M. BRE12-158: A Postneoadjuvant, Randomized Phase II Trial of Personalized Therapy Versus Treatment of Physician's Choice for Patients With Residual Triple-Negative Breast Cancer. J Clin Oncol. 2022 Feb 1;40(4):345-355. doi: 10.1200/JCO.21.01657. Epub 2021 Dec 15. PMID 34910554
- [Derived] Radovich M, Jiang G, Hancock BA, Chitambar C, Nanda R, Falkson C, Lynce FC, Gallagher C, Isaacs C, Blaya M, Paplomata E, Walling R, Daily K, Mahtani R, Thompson MA, Graham R, Cooper ME, Pavlick DC, Albacker LA, Gregg J, Solzak JP, Chen YH, Bales CL, Cantor E, Shen F, Storniolo AMV, Badve S, Ballinger TJ, Chang CL, Zhong Y, Savran C, Miller KD, Schneider BP. Association of Circulating Tumor DNA and Circulating Tumor Cells After Neoadjuvant Chemotherapy With Disease Recurrence in Patients With Triple-Negative Breast Cancer: Preplanned Secondary Analysis of the BRE12-158 Randomized Clinical Trial. JAMA Oncol. 2020 Sep 1;6(9):1410-1415. doi: 10.1001/jamaoncol.2020.2295. PMID 32644110
- See also: Hoosier Cancer Research Network Website — http://www.hoosiercancer.org

RESULTS

PARTICIPANT FLOW:
Period: Study Treatment
Arm/Group | Arm A (Genomically Directed Monotherapy) | Control Arm B (Observation/Standard Therapy)
Started | 71 | 122
Completed | 45 | 110
Not Completed | 26 | 12
Not completed — Disease Progression | 9 | 3
Not completed — Alternative therapy | 0 | 1
Not completed — No treatment, per protocol criteria | 0 | 4
Not completed — Patient Non compliance | 0 | 2
Not completed — Withdrawal by Subject | 5 | 2
Not completed — screen failure | 1 | 0
Not completed — AE/Side Effects/Complications | 8 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Disease Progression before treatment | 1 | 0
Not completed — Death | 1 | 0
Period: Follow up
Arm/Group | Arm A (Genomically Directed Monotherapy) | Control Arm B (Observation/Standard Therapy)
Started (Treatment and Follow up both are at different time period. Therefore, the number of subjects to start follow up is not equal to the number of subjects who have completed treatment.) | 70 | 122
Completed | 3 | 9
Not Completed | 67 | 113
Not completed — Lost to Follow-up | 4 | 9
Not completed — Refused to follow up | 5 | 4
Not completed — Death | 21 | 39
Not completed — study completed | 33 | 52
Not completed — screen failure | 2 | 0
Not completed — Pt. moved tx to Cancer Treatment Centers of America (Georgia). last contact was verbal on 3/10/16 | 0 | 1
Not completed — Disease progression - elected to participate in another clinical trial with no more follow up | 0 | 1
Not completed — Withdrawal by Subject | 2 | 2
Not completed — PI requested closure of site | 0 | 5

BASELINE CHARACTERISTICS:
Population: This population includes all subjects who were enrolled and found eligible and evaluable for this trial.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Genomically Directed Monotherapy) | Control Arm B (Observation/Standard Therapy) | Total
Number analyzed (Participants) | 71 | 122 | 193
Age, Customized [Count of Participants; unit: Participants]
  <= 45 | 29 | 40 | 69
  46-60 | 32 | 54 | 86
  61-75 | 10 | 27 | 37
  >= 76 | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71 | 122 | 193
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 14 | 17
  Not Hispanic or Latino | 66 | 106 | 172
  Unknown or Not Reported | 2 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 14 | 34 | 48
  White | 55 | 85 | 140
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
ECOG Performance Status [Count of Participants; unit: Participants] — Performance status are defined as follows :
  0 Fully active; no performance restrictions.
  1. Strenuous physical activity restricted; fully ambulatory and able to carry out light work.
  2. Capable of all self-care but unable to carry out any work activities. Up and about >50% of waking hours.
  3. Capable of only limited self-care; confined to bed or chair >50% of waking hours.
  4. Completely disabled; cannot carry out any self-care; totally confined to bed or chair.
  Participants
    0 | 60 | 100 | 160
    1 | 11 | 21 | 32
    2 | 0 | 1 | 1
Pathologic T stage at surgery [Count of Participants; unit: Participants] — Measure Description: Primary tumor (T) TX: Main tumor cannot be measured. T0: Main tumor cannot be found. T1, T2, T3, T4: Refers to the size and/or extent of the main tumor. The higher the number after the T, the larger the tumor or the more it has grown into nearby tissues. T's may be further divided to provide more detail, such as T3a and T3b.
  Participants
    T1 | 22 | 51 | 73
    T2 | 27 | 51 | 78
    T3 | 12 | 10 | 22
    T4 | 6 | 4 | 10
    Unknown | 4 | 6 | 10
Pathologic N stage at surgery [Count of Participants; unit: Participants] — Measure Description: Regional lymph nodes (N) NX: Cancer in nearby lymph nodes cannot be measured. N0: There is no cancer in nearby lymph nodes. N1, N2, N3: Refers to the number and location of lymph nodes that contain cancer. The higher the number after the N, the more lymph nodes that contain cancer.
  Participants
    N0 | 40 | 65 | 105
    N1 | 15 | 34 | 49
    N2 | 9 | 10 | 19
    N3 | 7 | 11 | 18
    Unknown | 0 | 2 | 2
M stage [Count of Participants; unit: Participants] — Measure Description: Distant metastasis (M) MX: Metastasis cannot be measured. M0: Cancer has not spread to other parts of the body. M1: Cancer has spread to other parts of the body.
  Participants
    M0 | 44 | 86 | 130
    Unknown | 27 | 36 | 63
Histologic grade [Count of Participants; unit: Participants] — Measure Description: Most tumors are graded as X, 1, 2, 3, or 4. Grade X: Grade cannot be assessed (undetermined grade) Grade 1: Well differentiated (low grade) Grade 2: Moderately differentiated (intermediate grade) Grade 3: Poorly differentiated (high grade) Grade 4: Undifferentiated (high grade)
  Participants
    1 | 0 | 1 | 1
    2 | 6 | 16 | 22
    3 | 64 | 102 | 166
    Unknown | 1 | 3 | 4
Lymph node involvement [Count of Participants; unit: Participants]
  Yes | 30 | 58 | 88
  No | 41 | 63 | 104
  Unknown | 0 | 1 | 1
RCB classsification [Count of Participants; unit: Participants] — Measure Description: RCB Classifications are defined as follows:
  I - minimal residual disease, II - moderate residual disease and III - extensive residual disease.
  Participants
    II | 33 | 54 | 87
    III | 14 | 22 | 36
    Unknown | 24 | 46 | 70

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Two-Year Disease-Free Survival (DFS)
Description: Two-year disease-free survival (DFS) in participants with confirmed triple negative breast cancer (TNBC) treated with a genomically directed therapy or standard of care following preoperative chemotherapy. The survival probabilities for arm A and arm B were estimated as 2 year disease free survival.
  DFS is defined as the duration of time from randomization to time of a DFS event, defined as local failure (invasive), regional failure, distant failure, contralateral breast cancer (invasive or non-invasive), or death from any cause.
Time Frame: From C1D1 until death or up to a maximum of 24 months.
Measure: Number; unit: percentage of participants
Arm/Group | Arm A (Genomically Directed Monotherapy) | Control Arm B (Observation/Standard Therapy)
Number analyzed (Participants) | 71 | 122
percentage of participants | 56.6 | 62.4

2. Secondary Outcome: Comparison Between Overall Disease-Free Survival
Description: Overall DFS in participants of arm A and B were compared with confirmed triple negative breast cancer (TNBC) treated with a genomically directed therapy or standard of care following preoperative chemotherapy.
  DFS is defined as the duration of time from randomization to time of a DFS event, defined as local failure (invasive), regional failure, distant failure, contralateral breast cancer (invasive or non-invasive), or death from any cause.
Time Frame: From C1D1 until death or up to a maximum of 58 months
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Arm A (Genomically Directed Monotherapy): Arm A : Genomically Directed Monotherapy: Participants randomized to Experimental Arm A will receive an FDA approved drug at standard dose for four cycles (12-16 weeks total duration, depending on cycle length). The CGTB will assign therapy to each participant individually based on biomarkers/pathways identified by DNA sequencing:
- Control Arm B (Observation/Standard Therapy): Arm B: Observation/Standard Therapy: Currently no standard therapy has proven efficacy in this patient population and thus observation alone would be considered standard of care. Additional therapy is permitted, however, if deemed appropriate by the treating physician.
Arm/Group | Arm A (Genomically Directed Monotherapy) | Control Arm B (Observation/Standard Therapy)
Number analyzed (Participants) | 71 | 122
months | NA [16.6 to NA] — Arm A did not drop to 50 % survival at the end of the available data, therefore neither the median nor upper limit could be calculated. | 48.7 [20.8 to NA] — Upper limit could not be reached since there weren't enough events at later times to get reliable upper CI for arm B.

3. Secondary Outcome: Comparison Between One Year Disease Free Survival
Description: One year DFS in participants of arm A and B were compared with confirmed triple negative breast cancer (TNBC) treated with a genomically directed therapy or standard of care following preoperative chemotherapy. The survival probabilities for arm A and arm B were estimated as 1 year disease free survival.
  Disease Free Survival is defined as the duration of time from randomization to time of a DFS event, defined as local failure (invasive), regional failure, distant failure, contralateral breast cancer (invasive or non-invasive), or death from any cause.
Time Frame: From C1D1 until death or up to a maximum of 12 months
Measure: Number; unit: percentage of participants
Arm/Group | Arm A (Genomically Directed Monotherapy) | Control Arm B (Observation/Standard Therapy)
Number analyzed (Participants) | 71 | 122
percentage of participants | 63.5 | 72.7

4. Secondary Outcome: Five-Year Overall Survival (OS) Rate
Description: 5-year overall survival (OS) in participants is determind with confirmed triple negative breast cancer (TNBC) treated with a genomically directed therapy or standard of care following preoperative chemotherapy. Here 5 - year survival probability to compare arms A and B has been reported.
  Overall Survival is defined as the time from start of treatment to death from any cause. Subjects who are alive are censored at their last visit dates.
Time Frame: From C1D1 until death or up to a maximum of 60 months
Measure: Number; unit: probability
Arm/Group | Arm A (Genomically Directed Monotherapy) | Control Arm B (Observation/Standard Therapy)
Number analyzed (Participants) | 71 | 122
probability | 0.52 | 0.62

5. Secondary Outcome: Number of Patients With Adverse Events as a Measure of Safety and Tolerability
Description: The safety and tolerability of the experimental arm A(genomically directed monotherapy) and control arm B(standard therapy) has been assessed using CTCAE v4.0. Number of subjects who had any adverse events or events greater than grade 3 were reported in this outcome measure.
Time Frame: From C1D1 until death or up to a maximum of 60 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Genomically Directed Monotherapy) | Control Arm B (Observation/Standard Therapy)
Number analyzed (Participants) | 71 | 122
Participants
  Number of patients had at least one adverse event of any grade | 65 | 34
  Number of patients had at least one grade 3 or greater adverse event | 23 | 10
  Number of patients had at least one grade 3 or greater treatment related adverse event | 23 | 10
  Number of patients having serious adverse event | 2 | 2

ADVERSE EVENTS:
Time Frame: From C1D1 up to at least 30 days after final protocol treatment or up to a maximum of 60 months.
Description: Adverse events will be recorded from the time of consent and for at least 30 days after final protocol treatment.
  SAEs must be reported during the course of the study within 24 hours of discovery of the event.
Arm/Group | Arm A (Genomically Directed Monotherapy) | Control Arm B (Observation/Standard Therapy)
All-Cause Mortality (participants affected / at risk) | 22/71 | 39/122
Serious Adverse Events (participants affected / at risk) | 2/71 | 2/122
Other Adverse Events (participants affected / at risk) | 65/71 | 33/122
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Genomically Directed Monotherapy) (N=71) | Control Arm B (Observation/Standard Therapy) (N=122)
BRACHIAL PLEXOPATHY (Nervous system disorders) | 1 (1) | 0 (0)
LUNG INFECTION (Infections and infestations) | 1 (1) | 0 (0)
MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDER - OTHER, SPECIFY (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
BREAST INFECTION (Infections and infestations) | 0 (0) | 1 (1)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS - OTHER, SPECIFY (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Genomically Directed Monotherapy) (N=71) | Control Arm B (Observation/Standard Therapy) (N=122)
ABDOMINAL PAIN (Gastrointestinal disorders) | 3 (3) | 4 (4)
AGITATION (Psychiatric disorders) | 1 (1) | 0 (0)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 2 (2) | 1 (2)
ALKALINE PHOSPHATASE INCREASED (Investigations) | 6 (7) | 0 (0)
ALLERGIC REACTION (Immune system disorders) | 1 (1) | 0 (0)
ALLERGIC RHINITIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
ALOPECIA (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
ANEMIA (Blood and lymphatic system disorders) | 6 (10) | 1 (1)
ANOREXIA (Metabolism and nutrition disorders) | 9 (12) | 0 (0)
ANXIETY (Psychiatric disorders) | 3 (3) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 8 (10) | 1 (1)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 4 (4) | 1 (2)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 13 (15) | 0 (0)
BLOOD BILIRUBIN INCREASED (Investigations) | 1 (1) | 0 (0)
BLURRED VISION (Eye disorders) | 3 (3) | 1 (1)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
BREAST INFECTION (Infections and infestations) | 2 (2) | 0 (0)
BREAST PAIN (Reproductive system and breast disorders) | 2 (2) | 2 (2)
CHEST WALL PAIN (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
CHOLECYSTITIS (Hepatobiliary disorders) | 1 (1) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 15 (19) | 0 (0)
COUGH (Respiratory, thoracic and mediastinal disorders) | 9 (11) | 0 (0)
CREATININE INCREASED (Investigations) | 2 (2) | 0 (0)
DEPRESSION (Psychiatric disorders) | 1 (1) | 0 (0)
DERMATITIS RADIATION (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
DIARRHEA (Gastrointestinal disorders) | 20 (32) | 8 (9)
DIZZINESS (Nervous system disorders) | 3 (3) | 1 (1)
DRY SKIN (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
DYSESTHESIA (Nervous system disorders) | 1 (1) | 0 (0)
DYSGEUSIA (Nervous system disorders) | 4 (5) | 1 (1)
DYSPEPSIA (Gastrointestinal disorders) | 5 (5) | 0 (0)
DYSPHAGIA (Gastrointestinal disorders) | 1 (1) | 0 (0)
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 10 (11) | 0 (0)
EDEMA FACE (General disorders) | 1 (1) | 0 (0)
EDEMA LIMBS (General disorders) | 2 (2) | 0 (0)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
FACIAL PAIN (General disorders) | 1 (1) | 0 (0)
FALL (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
FATIGUE (General disorders) | 36 (43) | 8 (8)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
FEVER (General disorders) | 1 (1) | 1 (1)
FLASHING LIGHTS (Eye disorders) | 1 (1) | 0 (0)
FLU LIKE SYMPTOMS (General disorders) | 2 (7) | 0 (0)
FLUSHING (Vascular disorders) | 1 (1) | 0 (0)
GASTROESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 2 (2) | 0 (0)
GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS (General disorders) | 1 (1) | 0 (0)
GENERALIZED MUSCLE WEAKNESS (Musculoskeletal and connective tissue disorders) | 1 (3) | 0 (0)
HEADACHE (Nervous system disorders) | 12 (15) | 1 (1)
HEMORRHOIDS (Gastrointestinal disorders) | 1 (1) | 0 (0)
HOARSENESS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
HOT FLASHES (Vascular disorders) | 4 (4) | 1 (1)
HYPERCALCEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 4 (6) | 1 (1)
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
HYPERTENSION (Vascular disorders) | 9 (11) | 7 (9)
HYPERTHYROIDISM (Endocrine disorders) | 1 (1) | 0 (0)
HYPOALBUMINEMIA (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
HYPOKALEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
HYPONATREMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
HYPOTHYROIDISM (Endocrine disorders) | 4 (5) | 0 (0)
INFECTIONS AND INFESTATIONS (Infections and infestations) | 2 (2) | 0 (0)
INSOMNIA (Psychiatric disorders) | 4 (4) | 1 (1)
IRRITABILITY (General disorders) | 1 (1) | 0 (0)
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
LOCALIZED EDEMA (General disorders) | 1 (1) | 0 (0)
LYMPHEDEMA (Vascular disorders) | 2 (2) | 0 (0)
LYMPHOCYTE COUNT DECREASED (Investigations) | 3 (3) | 1 (1)
MEMORY IMPAIRMENT (Nervous system disorders) | 1 (1) | 0 (0)
MUCOSAL INFECTION (Infections and infestations) | 1 (1) | 0 (0)
MUCOSITIS ORAL (Gastrointestinal disorders) | 5 (7) | 1 (1)
MUSCLE WEAKNESS TRUNK (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDER (Musculoskeletal and connective tissue disorders) | 3 (4) | 0 (0)
MYALGIA (Musculoskeletal and connective tissue disorders) | 5 (5) | 1 (1)
NAIL INFECTION (Infections and infestations) | 1 (2) | 1 (1)
NAIL LOSS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 23 (34) | 6 (6)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
NEOPLASMS BENIGN, MALIGNANT AND UNSPECIFIED (INCL CYSTS AND POLYPS) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
NEUTROPHIL COUNT DECREASED (Investigations) | 9 (12) | 0 (0)
ORAL DYSESTHESIA (Gastrointestinal disorders) | 1 (2) | 0 (0)
ORAL PAIN (Gastrointestinal disorders) | 2 (2) | 0 (0)
PAIN (General disorders) | 4 (5) | 0 (0)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 4 (6) | 0 (0)
PALMAR-PLANTAR ERYTHRODYSESTHESIA SYNDROME (Skin and subcutaneous tissue disorders) | 3 (5) | 6 (6)
PAPULOPUSTULAR RASH (Infections and infestations) | 1 (1) | 0 (0)
PARESTHESIA (Nervous system disorders) | 1 (1) | 0 (0)
PELVIC PAIN (Reproductive system and breast disorders) | 1 (1) | 1 (1)
PERIORBITAL EDEMA (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
PERIPHERAL MOTOR NEUROPATHY (Nervous system disorders) | 1 (1) | 0 (0)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 9 (10) | 2 (2)
PERSONALITY CHANGE (Psychiatric disorders) | 1 (1) | 0 (0)
PLATELET COUNT DECREASED (Investigations) | 6 (7) | 1 (1)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
PRESYNCOPE (Nervous system disorders) | 1 (2) | 0 (0)
PRURITUS (Skin and subcutaneous tissue disorders) | 4 (4) | 1 (1)
PSYCHIATRIC DISORDERS (Psychiatric disorders) | 1 (1) | 0 (0)
RASH ACNEIFORM (Skin and subcutaneous tissue disorders) | 6 (6) | 0 (0)
SINUS PAIN (Nervous system disorders) | 1 (1) | 0 (0)
SINUSITIS (Infections and infestations) | 1 (1) | 1 (1)
SKIN AND SUBCUTANEOUS TISSUE DISORDERS (Skin and subcutaneous tissue disorders) | 2 (3) | 1 (1)
SKIN INFECTION (Infections and infestations) | 2 (3) | 1 (1)
SKIN ULCERATION (Skin and subcutaneous tissue disorders) | 2 (4) | 0 (0)
SORE THROAT (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
SUPERFICIAL SOFT TISSUE FIBROSIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
TELANGIECTASIA (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
UPPER RESPIRATORY INFECTION (Infections and infestations) | 1 (1) | 2 (2)
URINARY TRACT INFECTION (Infections and infestations) | 3 (3) | 1 (1)
VAGINAL INFECTION (Infections and infestations) | 1 (1) | 0 (0)
VAGINAL INFLAMMATION (Reproductive system and breast disorders) | 1 (2) | 0 (0)
VOMITING (Gastrointestinal disorders) | 7 (8) | 1 (1)
WEIGHT GAIN (Investigations) | 2 (2) | 2 (2)
WEIGHT LOSS (Investigations) | 2 (3) | 0 (0)
WHITE BLOOD CELL DECREASED (Investigations) | 3 (3) | 1 (1)
WOUND DEHISCENCE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
BLOATING (Gastrointestinal disorders) | 0 (0) | 1 (1)
BLOOD AND LYMPHATIC SYSTEM DISORDERS (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
CARDIAC DISORDERS (Cardiac disorders) | 0 (0) | 1 (2)
DEHYDRATION (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
ENDOCRINE DISORDERS (Endocrine disorders) | 0 (0) | 1 (1)
ERYTHEMA MULTIFORME (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
FECAL INCONTINENCE (Gastrointestinal disorders) | 0 (0) | 1 (1)
GASTROINTESTINAL DISORDERS (Gastrointestinal disorders) | 0 (0) | 1 (1)
GASTROINTESTINAL PAIN (Gastrointestinal disorders) | 0 (0) | 1 (1)
GLUCOSE INTOLERANCE (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
HYPOTENSION (Vascular disorders) | 0 (0) | 1 (1)
PALPITATIONS (Cardiac disorders) | 0 (0) | 1 (1)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
SEROMA (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
SKIN HYPERPIGMENTATION (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-27): https://cdn.clinicaltrials.gov/large-docs/85/NCT02101385/Prot_SAP_000.pdf